CLINICAL TRIAL: NCT02943148
Title: Predictive Value of Striae Gravidarum Severity and Cesarean Scar Characteristics for Pelvic Adhesions at Repeat Cesarean Delivery
Brief Title: Prediction of Pelvic Adhesions at Repeat Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Other Study IDs: PACS
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Decrease Maternal Morbidity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Davey score for striae gravidarum

SUMMARY:
Several methods have been used to predict adhesions after abdominal operations. High-resolution ultrasonography, magnetic resonance imaging and scar healing properties were the methods that were evaluated in the English literature for this study. Estimating the likelihood of adhesions and related complications after prior surgery and assessing the severity of adhesion formation after surgery is not easy. Anticipating adhesions is very important to preventing complications by ensuring that the necessary preoperative preparations are in place and/or that appropriate cases are referred to a tertiary center.

ELIGIBILITY:
Inclusion Criteria:

1. Women with at least previous one cesarean
2. Full term (37- 41 weeks)
3. Women accepted to participate in the study

Exclusion Criteria:

1. History of pelvic inflammatory disease
2. History of endometriosis
3. Previous pelvic surgery other than cesarean
4. History of wound site infections
5. History of long corticosteroid use
6. Women with midline incisions
7. Women with placenta accreta
8. Women refuse to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Women who will be admitted to our Labor Ward for emergency or elective cesarean section will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Rate of of abdominal adhesions in relation to striae scoring system | 30 min

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes